CLINICAL TRIAL: NCT03290638
Title: Comparison of Dehydrated Human Amnion-Chorion and Type 1 Bovine Collagen Membranes for Guided Bone Regeneration (Socket Augmentation) : A Clinical and Histological Study
Brief Title: Comparison of Dehydrated Human Amnion-Chorion and Type 1 Bovine Collagen Membranes for Guided Bone Regeneration
Acronym: GBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samer Faraj (Other)
Responsible Party: Sponsor-Investigator, Samer Faraj, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13-0540-F3R
Record Dates: First submitted 2017-09-06; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Ridge Deficiency
Keywords: Guided Bone Regeneration; Dehydrated Human Amnion Chorion Membrane; Type I Bovine Collagen Membrane; Ridge Preservation; Ridge Healing; Teeth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dehydrated Human Amnion Chorion Membrane (Experimental): This membrane was investigated to evaluate its use as an open barrier for guided bone regeneration (GBR) after tooth extraction and to determine whether intentional exposure of this membrane to the oral environment compromises ridge dimensions and bone vitality for implant placement.
  Interventions: Procedure: Guided Bone Regeneration (GBR)
- Type I Bovine Collagen Membrane (Active Comparator): This membrane has been tested as an open barrier for GBR after tooth extraction. The intentional use of this membrane to the oral environment did not compromise ridge dimensions and bone vitality for implant placement.
  Interventions: Procedure: Guided Bone Regeneration (GBR)

INTERVENTIONS:
Procedure: Guided Bone Regeneration (GBR) — Teeth Extraction With Bone Grafting and Membrane
  Other Names: Ridge Preservation

SUMMARY:
The objective of this randomized clinical study was to evaluate the use of dehydrated human amnion-chorion membrane as an exposed barrier for guided bone regeneration (GBR) after tooth extraction and to determine whether intentional exposure of this membrane to the oral environment compromises ridge dimensions and bone vitality for implant placement.

DETAILED DESCRIPTION:
Forty-three patients requiring extraction of at least one tooth and delayed implant placement were randomly assigned to either an experimental or a control group. For both groups, demineralized freeze-dried bone allograft was used to graft the socket. For the control group, Type I bovine collagen was used as a membrane; for the experimental group, human amnion-chorion membrane was used. For both groups, the barrier membranes were left exposed, and no primary closure was achieved. Patients returned for implant placement after a mean healing period of 19.5 weeks, at which time a core bone biopsy specimen 2 mm in diameter was obtained for histomorphometric analyses. Clinical ridge dimensions were measured at the times of extraction and implant placement.

ELIGIBILITY:
Inclusion Criteria: .

Patients included in the study were required:

* Not to be completely edentulous.
* To have at least 1 tooth that could not be saved and for which extraction and delayed implant placement were planned

Exclusion Criteria: Patients were excluded if they :

* Had received radiation therapy
* Were taking antiresorptive medication (i.e., bisphosphonate or denosumab)
* Had uncontrolled systemic disorders (such as uncontrolled diabetes, congestive heart failure, or acute odontogenic infections)
* Were smokers (more than 10 cigarettes per day)
* Were pregnant or breastfeeding.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Ridge Dimensional Changes | Alveolar Ridge Dimensional Changes were taken at the extraction time and at the time of implant placement. Mean = 19.5 weeks
  Clinical ridge height changes were taken with a thermoplastic triad stent, and a University of North Carolina (UNC) 15 periodontal probe. Ridge width changes measurements were taken with a metal bone caliper. Alveolar ridge dimensional changes in height and width were measured at the times of extraction and at the time of implant placement.
Alveolar Ridge Bone Vitality | Mean= 19.5 weeks after tooth extraction and bone grafting
  a core bone biopsy specimen 2 mm in diameter was obtained from the center of the root at the time of implant placement for histomorphometric analyses

SECONDARY OUTCOMES:
Ridge Healing Evaluation | Two weeks form the time of the extraction
  Pictures of the healing ridges were taken using clinical macro lens photography